CLINICAL TRIAL: NCT00982124
Title: An International, Multicenter, Open-label, Efficacy and Safety Trial of Intravenous Zoledronic Acid in Infants Less Than One Year of Age, With Severe Osteogenesis Imperfecta
Brief Title: An Efficacy and Safety Trial of Intravenous Zoledronic Acid in Infants Less Than One Year of Age, With Severe Osteogenesis Imperfecta
Acronym: INFOI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Francis H. Glorieux, Principal Investigator, Shriners Hospitals for Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SHC-INFOI; IRB - A06-M73-06A; Health Canada - 9427-S1926-24C
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta; Infants with moderate to severe Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Zoledronic Acid

ARMS (1):
- Treatment Arm (only) (Experimental): Zoledronic acid infusion
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — Each patient is to receive an initial dose of zoledronic acid of 0.0125 mg per kg body weight, then subsequent doses of zoledronic acid at a dose of 0.025 mg per kg body weight once every 12 to 13 weeks for 104 weeks (total of 8 doses).
  Other Names: Aclasta

SUMMARY:
The investigators have currently finished conducting an international multi-center trial that compares the efficacy and safety of pamidronate and zoledronate in the treatment of moderate to severe forms of Osteogenesis Imperfecta (OI). This trial has included only children above one year of age. The aim of the current study is to extend the observations of that currently finished study to infants below 1 year of age. Moreover, it is possible to administer zoledronate in a single short infusion instead of the three-day cycles with Pamidronate, therefore decreasing patient and family burdens with shorter stays in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Children, male or female 2 weeks to < 12 months of age, at least at 38 weeks gestational age.
* Any child with phenotypic OI type II, III or IV.
* Any child classified as OI type I, V-VIII that has had at least two or more previous fractures of long bone, or vertebral compression fractures, and a low bone mineral density.
* No previous treatment with bisphosphonates.
* Negative urine protein as measured by dipstick. One repeat assessment of the urine protein will be allowed.

Exclusion Criteria:

* Blood oxygen saturation of less than 90% in room air.
* Serum creatinine level greater than 56 µmol/L.
* Any clinically significant clinical laboratory abnormalities at screening.
* Treatment with any investigational drug within the past 30 days.
* Patients who are unlikely to be able to complete the study or comply with the visit schedule.
* Any disease or planned therapy which will interfere with the procedures or data collection of this trial.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2007-10; Primary Completion 2015-09 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial is to assess the change in lumbar spine bone mineral density Z-score at month 24 relative to baseline in zoledronic acid treated infants compared to historical controls. | 3 times during 10 visits within 2 years

SECONDARY OUTCOMES:
To assess the effect of zoledronic acid on the number of clinical fractures &/or vertebral compressions that occur over a two year period compared to untreated historical controls in infants. | 3 times during 10 visits within 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Francis H. Glorieux, MD, PhD, Principal Investigator — McGill University
Locations (1):
- Shriners Hospital for Children, Montreal, Quebec, Canada